CLINICAL TRIAL: NCT05652972
Title: KETO-MINOX: The Effect of Isocaloric, Energy-restrictive, KETOgenic Diet on Metabolism, Inflammation, Nutrition Deficiencies and OXidative Stress in Women With Overweight and Obesity
Brief Title: Effect of KETOgenic Diet on Metabolism, Inflammation, Nutrition Deficiencies and OXidative Stress in Women With Overweight
Acronym: KETO-MINOX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Academy of Sciences (Other)
Collaborators: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Natalia Drabińska, Principal Investigator, Polish Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/41/B/NZ9/01278
Record Dates: First submitted 2022-11-29; First posted 2022-12-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Overweight and Obesity
Keywords: diet; nutrition; ketogenic diet; inflammation; oxidative stress; overweight
MeSH Terms: conditions — Overweight; Obesity; Inflammation | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Experimental): 40 women which will follow the ketogenic diet with 1700 kcal daily for 8 weeks
  Interventions: Other: Ketogenic diet
- Control diet (Active Comparator): 40 women which will follow the standard diet with 1700 kcal daily for 8 weeks
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Ketogenic diet — 1700 kcal ketogenic diet (fat: protein: carbohydrate ratio of 70:20:10)
  Arms: Ketogenic diet
Other: Control diet — 1700 kcal standard diet (fat: protein: carbohydrate ratio of 20:30:50)
  Arms: Control diet

SUMMARY:
In recent times, the prevalence of obesity increases, reaching an epidemic scale. Elevated body weight is a risk factor in the development of several diseases such as diabetes, hypertension and cancer. Therefore, obesity management solutions, such as diet therapy are needed. The key issue is to choose the most appropriate diet to obtain an efficient outcome in losing weight, without experiencing adverse effects and a decrease in general health. A ketogenic diet, an auxiliary therapy for epilepsy, is recently one of the options commonly used for losing weight by overweight individuals, tempted by the commercials and internet influencers. However, there is limited knowledge about the effect of this diet on human health. To date, the majority of studies were conducted with a very-low-calorie regime applied before the bariatric surgeries, which itself may affect the loss of body weight, and in most studies, the control diets were missing. Taking into consideration that a ketogenic diet is an extremely eliminating diet, there is a risk of nutritional deficiencies after following it. Therefore, there is a strong need for more in-depth and comprehensive elucidation of the safety and physiological effects of the ketogenic diet used for the weight loss in overweight and obese individuals.

This Project aims to evaluate the effectiveness of the eight-week, isocaloric, energy-restricted, ketogenic diet as a weight management solution in women with overweight and obesity compared to the standard, balanced diet with the same calorie content.

DETAILED DESCRIPTION:
In recent times, the prevalence of obesity increases, reaching an epidemic scale. A new factor supporting a weight gain is a current coronaviros (COVID-19) pandemic, associated with reduced physical activity, high stress and overeating, which resulted in 2-5 kg weight gain in 20 % of the American population within a few months 1. Elevated body weight is a risk factor in developing several diseases such as diabetes, hypertension and cancer. Therefore, obesity management solutions, such as diet therapy, are needed. The critical issue is to choose the most appropriate diet to obtain an efficient outcome in losing weight without experiencing adverse effects and a decrease in general health. A ketogenic diet, an auxiliary therapy for epilepsy, is recently one of the options commonly used for losing weight by individuals with overweight, tempted by the commercials and internet influencers. However, there is limited knowledge about the effect of this diet on human health. To date, the majority of studies were conducted with a very low-calorie regime applied before the bariatric surgeries, which itself may affect the loss of body weight. In most studies, the control diets were missing. Considering that a ketogenic diet is an extremely eliminating diet, there is a risk of nutritional deficiencies after following it. Therefore, there is a strong need for more in-depth and comprehensive elucidation of the safety and physiological effects of the energy-restricted ketogenic diet used for weight loss in individuals with overweight and obese.

This Project aims to evaluate the effectiveness of the eight-week, isocaloric, energy-restricted, ketogenic diet as a weight management solution in women with overweight and obesity compared to the standard, balanced diet with the same calorie content.

ELIGIBILITY:
Inclusion Criteria:

* women
* age 18-45
* overweight (BMI 27 - 35)
* motivation to lose weight and participate in the nutritional intervention trial

Exclusion Criteria:

* overweight/obesity secondary to genetic syndromes
* endocrine diseases, acute systemic disease, autoimmune disorders
* pregnancy
* breastfeeding
* type 1 and 2 diabetes
* any other chronic diseases requiring pharmacotherapy (including topical steroids in allergy disorders
* supplement or medication use influencing appetite, weight or metabolism)
* participation in other clinical trials
* severe obesity (BMI > 35)
* > 3 kg weight loss 12 weeks before the initial test day
* extreme changes in exercise intensity 4 weeks prior
* any diagnosed psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers (G-CSF, GM-CSF, INF-gamma, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17, MCP-1, MIP-1b, TNF-a) | 12 months
  Analysis using Bio-Plex Pro™ Human Cytokine 17-plex Assay in serum.
Oxidative stress markers | 12 months
  analysis of malondialdehyde, superoxide dismutase, 8-isoprostane and 8-hydroxydeoxyguanosine (8-OHdG) using commercial ELISA kits in serum.

SECONDARY OUTCOMES:
Body weight and composition | 12 months
  Body weight in kg and composition in % will be measured using Body Composition Analyser
Waist circumference | 12 months
  The waist circumference in cm will be measured using a standard measurement tape.
Free amino acids | 12 months
  Analysis of free amino acids in serum using gas chromatography-mass spectrometry, expressed in nmol/mL
Fat-soluble vitamins | 12 months
  Fat-soluble vitamins in serum using commercial ELISA kits (vitamin D) and high-performance liquid chromatography (vitamin A,E & K)
Metabolites in breath | 12 months
  Volatile organic compounds in breath will be measured using dwo dimensional chromatography with time of flight mass spectrometry (GCxGC-ToFMS)
Obesity-related markers (C-peptide, ghrelin, gastric inhibitory peptide (GIP), glucagon-like peptide 1 (GLP-1), glucagon, insulin, leptin, plasminogen activation inhibitor-1 (PAI-1), resistin and visfatin, adipsin and adiponectin) | 12 months
  Analyses will be performed using Bio-Plex Assays

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Drabińska, PhD, Principal Investigator — Institute of Animal Reproduction and Food Reseach, Polish Academy of Sciences in Olsztyn; Jerzy Romaszko, MD, PhD, Principal Investigator — Deaprtment of Family Medicine and Infectious Diseases, Faculty of Medical Sciences, University of Warmia and Mazury
Locations (2):
- Poland (2):
  - Department of Family Medicine and Infectious Diseases, Faculty of Medical Sciences, University of Warmia and Mazury, Olsztyn
  - Institute of Animal Reproduction and Food Research, Polish Academy of Sciences, Olsztyn

IPD SHARING:
Plan to Share IPD: Yes
During the project only new data will be acquired and/or generated. No existing data re-usage is planned. Similar data do not exist yet, thus the planned project will be the only source/origin of them.
  In the project the following data will be generated: numerical data, texts and graphical data (chromatography).
  During the the project, two types of data will be generated to further processing:
  1. automatic measurement data resulting from the equipment, obtained using the validated methodologies and calibrated equipments with the predefined replicates.
  2. non-automatic measurement data resulting from carried out experiments - data documented manually and then entered into a spreadsheets and obtained after the statistical evaluation.
  All data will be successfully published in prestigious journals with high Impact Factor. Thus, they will be evaluated by the expert reviewers in the process of revision.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Drabinska N, Romaszko J, White P. The effect of isocaloric, energy-restrictive, KETOgenic diet on metabolism, inflammation, nutrition deficiencies and oxidative stress in women with overweight and obesity (KETO-MINOX): Study protocol. PLoS One. 2023 May 8;18(5):e0285283. doi: 10.1371/journal.pone.0285283. eCollection 2023. PMID 37155645